CLINICAL TRIAL: NCT03773471
Title: A Multi-Center Cluster Randomized Controlled Clinical Trial to Determine the Impact of a Mobile Health Application on Rheumatoid Arthritis Shared Decision Making
Brief Title: A Multi-Center Clinical Trial to Determine the Impact of a Mobile Health Application on Rheumatoid Arthritis Shared Decision Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John M. Davis, III, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-005947
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Standard of care
- Intervention Arm (Experimental): Mobile Health App
  Interventions: Behavioral: Mobile Health App

INTERVENTIONS:
Behavioral: Mobile Health App — ArthritisPower App
  Arms: Intervention Arm

SUMMARY:
The overall goal is to improve shared decision-making (SDM) about treatment options and thereby enhance disease outcomes and health-related quality of life (HRQOL) for patients with rheumatoid arthritis (RA). The objective of this study is to engage patients in using the ArthritisPower application on a weekly basis during the time between clinic appointments for collection of data on self-reported disease activity and patient-reported outcomes (PROs), and to display the data using an iPad to the patients and their rheumatology health care providers (HCPs) at the point of care for SDM.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 18 years.
2. Fulfillment of the ACR/EULAR 2010 classification criteria for RA [9].
3. Moderate or high disease activity, according to CDAI ≥ 10, at the baseline visit.
4. Intent to modify DMARD therapy (i.e., adding a DMARD, switching to a new DMARD, or changing DMARD dosage) by the patient and HCP.

Exclusion criteria:

1. Current or previous use of ArthritisPower™ by the patient.
2. Lack of access to an ArthritisPower™ compatible device (e.g., smartphone, tablet, or computer)
3. Inability or unwillingness to participate with using the ArthritisPower™ app for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
- Determine the impact of ArthritisPower™ integration into the clinical evaluation of patients with RA on the primary endpoint of clinical improvement as defined by the continuous change in the Clinical Disease Activity Index (CDAI) (1). | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: John M Davis, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Michigan Medicine - Rheumatology, Ann Arbor, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials